CLINICAL TRIAL: NCT01516476
Title: A Multi-Center, Double-Blind, Randomized, Placebo-Controlled, Parallel-Group Study to Assess the Efficacy and Safety of RO6807952 in Type 2 Diabetic Patients Inadequately Controlled With Metformin Alone
Brief Title: Study of RO6807952 in Patients With Diabetes Mellitus Type 2
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BP27804
Record Dates: First submitted 2012-01-12; First posted 2012-01-24 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Liraglutide Arm (Experimental)
  Interventions: Drug: liraglutide
- Placebo Arm (Placebo Comparator)
  Interventions: Drug: Placebo
- RO6807952 Arm 1 (Experimental)
  Interventions: Drug: RO6807952
- RO6807952 Arm 2 (Experimental)
  Interventions: Drug: RO6807952

INTERVENTIONS:
Drug: Placebo — Placebo for 12 weeks
  Arms: Placebo Arm
Drug: RO6807952 — multiple doses for 12 weeks
  Arms: RO6807952 Arm 1
Drug: RO6807952 — multiple doses for 12 weeks
  Arms: RO6807952 Arm 2
Drug: liraglutide — liraglutide for 12 weeks
  Arms: Liraglutide Arm

SUMMARY:
This randomized, double-blind, placebo-controlled, multi-center study will evaluate the efficacy and safety of RO6807952 in patients with diabetes mellitus type 2 inadequately controlled with metformin alone. Patients will be randomized to receive doses of RO6807952, placebo, or liraglutide. The anticipated time on study treatment is 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients >/= 18 and </=70 years of age
* Diagnosis of diabetes mellitus, type 2 for at least 3 months
* Treated with a stable dose of metformin
* Hemoglobin A1c >/=7.0% and </=10.5% at screening
* Fasting plasma glucose </=240 mg/dL at screening
* Body mass index >/=27 kg/m2 and </=42 kg/m2 at screening
* Willing and able to maintain existing diet and exercise habits throughout the study
* C-peptide >1.5 ng/mL at screening

Exclusion Criteria:

* History of significant liver or kidney disease
* History of uncontrolled hypertension
* History of significant cardiovascular disease
* History of significant diabetic complications
* History of significant gastrointestinal conditions
* History of weight loss surgery or procedures involving the gastrointestinal tract
* History of chronic or acute pancreatitis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2011-11; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Change in hemoglobin A1c (HA1c) | Baseline and 12 weeks

SECONDARY OUTCOMES:
Change in fasting plasma glucose | Baseline and 12 weeks
Safety (incidence of adverse events) | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Cincinnati, Ohio, United States